CLINICAL TRIAL: NCT07171684
Title: Single vs Multi-Dose Insulin for Glycemic Control (SUGAR): A Randomized Noninferiority Trial
Brief Title: Single vs Multi-Dose Insulin for Glycemic Control (SUGAR)
Acronym: SUGAR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Emily B. Rosenfeld, DO, Principal Investigator, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro2025001063
Record Dates: First submitted 2025-08-30; First posted 2025-09-12 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-09

CONDITIONS: Diabetes in Pregnancy; Gestational Diabetes
Keywords: insulin glargine; insulin lispro; gestational diabetes; diabetes; pregnancy; noninferiority
MeSH Terms: conditions — Diabetes, Gestational; Diabetes Mellitus | interventions — Insulin Glargine; Insulin Lispro

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Insulin glargine alone (Experimental): Once daily dosing of insulin glargine
  Interventions: Drug: Insulin glargine alone
- Insulin glargine + Insulin lispro (Active Comparator): Once daily dosing of insulin glargine plus three times per day dosing of insulin lispro with each meal
  Interventions: Drug: Insulin glargine + insulin lispro

INTERVENTIONS:
Drug: Insulin glargine alone — Once daily dosing of insulin glargine
  Arms: Insulin glargine alone
Drug: Insulin glargine + insulin lispro — Once daily dosing of insulin glargine + three times daily dosing of insulin lispro with meals
  Arms: Insulin glargine + Insulin lispro

SUMMARY:
The goal of this clinical trial is to see if diabetes in pregnancy can be treated with once daily dosing of insulin instead of once daily dosing plus insulin with meals. The main question this study aims to answer is:

1. Can a once daily dose of long-acting insulin control blood sugars as well as long-acting insulin plus meal-time insulin?
2. Do babies born to mothers who take one dose of long-acting insulin have more complications after birth than babies born to mothers who take long-acting and meal-time insulin? Researchers will compare one dose of long-acting insulin per day to this plus three doses of short-acting insulin with each meal to see if blood sugars are controlled.

Participants will send their blood sugar logs to the study staff weekly, instead of to their OB/GYN, for adjustments to their insulin dosing.

DETAILED DESCRIPTION:
Purpose/Specific Aims

The purpose of this study is to determine if a single dose of long-acting insulin is non-inferior to long-acting insulin plus prandial insulin to manage diabetes in pregnancy, measured by a composite neonatal outcome of NICU admission, neonatal hyperglycemia, neonatal hypoglycemia, large for gestational age, shoulder dystocia, hyperbilirubinemia, stillbirth, and neonatal death.

A. Objectives:

This study aims to compare neonatal outcomes of patients with diabetes in pregnancy to determine if a single dose of long-acting insulin is non-inferior to long-acting insulin plus prandial insulin.

B. Hypotheses / Research Question(s):

The hypothesis is that once-daily long-acting insulin glargine is noninferior to long-acting insulin glargine in combination with prandial short-acting insulin lispro, which is the current standard of care at our institution, for glycemic management of gestational diabetes mellitus and type 2 diabetes mellitus in pregnancy, as measured by a composite neonatal outcome. The composite outcome includes NICU admission, neonatal hyperglycemia, neonatal hypoglycemia, large for gestational age, shoulder dystocia, hyperbilirubinemia stillbirth, and neonatal death, which are associated with inadequate glycemic management during pregnancy.

Research Procedure:

Individuals will be recruited for the study during routine prenatal care visits or during initial, standard of care consults with Robert Wood Johnson Maternal Fetal Medicine Specialists when insulin use is suggested for glycemic management. Gestational age at enrollment will vary from patient to patient, but all patients will be enrolled when insulin is clinically indicated to manage their diabetes. If patients choose to participate in the study, they will be randomized to standard of care (long-acting insulin glargine plus prandial insulin lispro) or the experimental group (long-acting insulin glargine only). This study is a noninferiority study between standard of care dosing strategies. This question is best investigated via a noninferiority design, given the potential to improve the currently accepted treatment by reducing patient burden. During this initial consult, a review of medical records is completed, regardless of study participation.

After randomization, both groups will receive dosing instructions per the Insulin Dosing Algorithm. The study utilizes a similar process to the MFM clinical workflow. Patients test their blood glucose at home, and send their blood glucose logs to MFM nurse or study team member, which includes an MFM fellow. If insulin dose adjustments are needed due to hyper- or hypoglycemia, these dose modifications will be made based off the Insulin Dosing Algorithm (Figure 1), and be recorded in the Insulin Dosing Log and communicated with the patients.

Patients will remain in their randomized group unless participation in the experimental group with insulin glargine alone is not sufficient to achieve glycemic targets, as evidenced by three dose increases with persistent hyperglycemia. In that case, patients revert to standard of care group but remain in the study.

The final study procedure is data abstraction and survey administration following childbirth. The Delivery Outcomes form on REDCap will be utilized to abstract relevant maternal and neonatal outcomes from the labor and delivery hospitalization, as well as any hospitalizations indicative of maternal complications prior to childbirth. Finally, the Diabetes Treatment and Satisfaction Questionnaire - Status (DTSQs) will be administered around the time of delivery, optimally at 38 weeks gestation to assess differences in perspective based on frequency of insulin injection between the two groups. This survey has been well-validated for assessing patient satisfaction with insulin treatment. Importantly, the DTSQs is appropriately sensitive to detect changes based on this study's independent variable, as it has been used in a similar study to analyze satisfaction changes in standard insulin versus analogue insulins, as well as changes in long-term and short-term insulin. Study participation ends with the completion of the DTSQs.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 2 diabetes mellitus or A2 gestational diabetes mellitus requiring insulin use during pregnancy
* Aged between 18-50
* Speak English or Spanish

Exclusion Criteria:

* Pre-existing use of insulin
* Gestational Age > or = 35w0d
* Planning to follow-up with a doctor not associated with RWJ Barnabas and/or deliver at a hospital other than RWJUH
* Unwilling or unable to upload or email weekly blood sugar logs
* Contraindication to Lispro or Lantus insulin, or patient chooses to not utilize insulin therapy
* Fetal anomaly present

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 176 (Estimated)
Dates: Start 2025-11-26 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-05-15 (Estimated)

PRIMARY OUTCOMES:
Composite outcome | From enrollment to delivery
  NICU admission, neonatal hyperglycemia, neonatal hypoglycemia, large for gestational age, shoulder dystocia, hyperbilirubinemia stillbirth, and neonatal death

SECONDARY OUTCOMES:
Compliance with medication | From enrollment to delivery
  How often participant is taking the prescribed insulin regimen
% of patients in experimental group who are able to remain on insulin glargine only | From enrollment to delivery
  Percentage of patients who remain on insulin glargine only throughout their pregnancy instead of switching to standard of care due to uncontrolled blood sugars
Maternal complication rates | From enrollment to maternal discharge from delivery hospitalization
  Maternal complications include cesarean section, hypertensive disorders of pregnancy, use of insulin during labor, pre-eclampsia, number of days spent in hospital
Birth complications | Delivery to discharge of infant from birth hospitalization
  Pre-term delivery, shoulder dystocia, stillbirth rate. All will be reported as yes/no
Neonatal complications | Delivery to discharge during birth hospitalization
  Temperature regulation issues, polycythemia vera, admission to NICU. All will be measured as yes/no
Birthweight | Delivery, first weight recorded
  Neonatal birthweight in grams
APGAR Scores | Delivery to 5 minutes after delivery
  APGAR score at 1 and 5 minutes after delivery
Neonatal hospital stay | Delivery of neonate to discharge from birth hospitalization
  Number of days the neonate is admitted to the hospital during birth hospitalization
Patient satisfaction | From enrollment to delivery
  Patient satisfaction with randomized treatment group, as assessed through Diabetes Treatment Satisfaction Questionnaire.
  Treatment Satisfaction scale total has a minimum of 0 and a maximum of 36. A score of 36 indicates a patient is very satisfied with their treatment and a score of 0 indicates a patient is very unsatisfied with their treatment. Perceived frequency of hyperglycemia (item 2) and perceived frequency of hypoglycemia (item 3) are treated individually in data analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Emily Rosenfeld, DO, Principal Investigator — Rutgers Robert Wood Johnson Medical School
Locations (1):
- Robert Wood Johnson Univeristy Hospital, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bradley C, Lewis KS. Measures of psychological well-being and treatment satisfaction developed from the responses of people with tablet-treated diabetes. Diabet Med. 1990 Jun;7(5):445-51. doi: 10.1111/j.1464-5491.1990.tb01421.x. PMID 2142043
- [Background] Senat MV, Affres H, Letourneau A, Coustols-Valat M, Cazaubiel M, Legardeur H, Jacquier JF, Bourcigaux N, Simon E, Rod A, Heron I, Castera V, Sentilhes L, Bretelle F, Rolland C, Morin M, Deruelle P, De Carne C, Maillot F, Beucher G, Verspyck E, Desbriere R, Laboureau S, Mitanchez D, Bouyer J; Groupe de Recherche en Obstetrique et Gynecologie (GROG). Effect of Glyburide vs Subcutaneous Insulin on Perinatal Complications Among Women With Gestational Diabetes: A Randomized Clinical Trial. JAMA. 2018 May 1;319(17):1773-1780. doi: 10.1001/jama.2018.4072. PMID 29715355
- [Background] Figueroa Gray M, Hsu C, Kiel L, Dublin S. "It's a Very Big Burden on Me": Women's Experiences Using Insulin for Gestational Diabetes. Matern Child Health J. 2017 Aug;21(8):1678-1685. doi: 10.1007/s10995-017-2261-8. PMID 28092062
- [Background] Hartling L, Dryden DM, Guthrie A, Muise M, Vandermeer B, Donovan L. Benefits and harms of treating gestational diabetes mellitus: a systematic review and meta-analysis for the U.S. Preventive Services Task Force and the National Institutes of Health Office of Medical Applications of Research. Ann Intern Med. 2013 Jul 16;159(2):123-9. doi: 10.7326/0003-4819-159-2-201307160-00661. PMID 23712381
- [Background] Crowther CA, Hiller JE, Moss JR, McPhee AJ, Jeffries WS, Robinson JS; Australian Carbohydrate Intolerance Study in Pregnant Women (ACHOIS) Trial Group. Effect of treatment of gestational diabetes mellitus on pregnancy outcomes. N Engl J Med. 2005 Jun 16;352(24):2477-86. doi: 10.1056/NEJMoa042973. Epub 2005 Jun 12. PMID 15951574
- [Background] Scholtens DM, Kuang A, Lowe LP, Hamilton J, Lawrence JM, Lebenthal Y, Brickman WJ, Clayton P, Ma RC, McCance D, Tam WH, Catalano PM, Linder B, Dyer AR, Lowe WL Jr, Metzger BE; HAPO Follow-up Study Cooperative Research Group; HAPO Follow-Up Study Cooperative Research Group. Hyperglycemia and Adverse Pregnancy Outcome Follow-up Study (HAPO FUS): Maternal Glycemia and Childhood Glucose Metabolism. Diabetes Care. 2019 Mar;42(3):381-392. doi: 10.2337/dc18-2021. Epub 2019 Jan 7. PMID 30617141
- [Background] HAPO Study Cooperative Research Group. Hyperglycemia and Adverse Pregnancy Outcome (HAPO) Study: associations with neonatal anthropometrics. Diabetes. 2009 Feb;58(2):453-9. doi: 10.2337/db08-1112. Epub 2008 Nov 14. PMID 19011170
- [Background] Ainuddin JA, Karim N, Zaheer S, Ali SS, Hasan AA. Metformin treatment in type 2 diabetes in pregnancy: an active controlled, parallel-group, randomized, open label study in patients with type 2 diabetes in pregnancy. J Diabetes Res. 2015;2015:325851. doi: 10.1155/2015/325851. Epub 2015 Mar 22. PMID 25874236
- [Background] Hickman MA, McBride R, Boggess KA, Strauss R. Metformin compared with insulin in the treatment of pregnant women with overt diabetes: a randomized controlled trial. Am J Perinatol. 2013 Jun;30(6):483-90. doi: 10.1055/s-0032-1326994. Epub 2012 Oct 24. PMID 23096052
- [Background] Lain KY, Catalano PM. Metabolic changes in pregnancy. Clin Obstet Gynecol. 2007 Dec;50(4):938-48. doi: 10.1097/GRF.0b013e31815a5494. PMID 17982337
- [Background] American Diabetes Association Professional Practice Committee. 15. Management of Diabetes in Pregnancy: Standards of Care in Diabetes-2024. Diabetes Care. 2024 Jan 1;47(Suppl 1):S282-S294. doi: 10.2337/dc24-S015. PMID 38078583